CLINICAL TRIAL: NCT01195740
Title: Family Therapy as Hospital Aftercare for Adolescent Suicide Attempters
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-006296
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Suicide Ideation; Depression; Family Conflict
Keywords: Suicide Ideation; Depression; Family Conflict
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attachment Based Family Therapy (Experimental)
  Interventions: Behavioral: Attachment Based Family Therapy
- Enhanced Usual Care (Active Comparator)
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Attachment Based Family Therapy — ABFT has three phases. In phase one, treatment focuses on helping the adolescent identify past and present family conflicts that have strained the attachment bond and damaged trust. Adolescents and parents are taught new communication and affect regulation skills in preparation for reparative conversations in phase two. This phase of treatment involves adolescents and parents discussing these past and present conflicts using their new communication skills. The final phase of treatment focuses on promoting adolescent autonomy (i.e., improving school productivity, finding a job, etc.). For the suicidal/depressed adolescent, this can decrease isolation and increase exposure to positive experiences. To accomplish these goals, there are five ABFT treatment tasks. Each task may take one or several sessions. Youth randomized to this condition will receive approximately 14 weeks of ABFT. One orientation meeting will occur, whenever possible, on the inpatient unit prior to discharge.
  Other Names: Attached Based Family Therapy; ABFT
  Arms: Attachment Based Family Therapy
Behavioral: Enhanced Usual Care — Belmont offers the Therapeutic Bridge Program, funded by the Pew Charitable Trusts, which helps adolescents make the transition from the hospital back to home, school and community behavioral health services. The program serves as a "bridge" between inpatient and outpatient care during the first 90 days after discharge, linking them to supportive services. Aftercare begins at the point of intake. Several discharge planning meetings are held with the adolescent and parents during the inpatient stay. The range of services are based on the patient and families' need, and may include meeting with school personnel , conducting home visits or making referrals to other community services agencies. The main objective is to secure outpatient mental health services for the patient. These services will be enhanced by the weekly research tracking, assessment and 24-hour crisis phone line which will call into a cell phone rotated among the licensed mental health professionals on the research team.
  Arms: Enhanced Usual Care

SUMMARY:
Few empirically-based treatment models exist for adolescent suicide attempters post psychiatric hospitalization, despite the fact that managed care has limited the role of hospitalization to stabilization, rather than remission. This study will test the efficacy and initial outcomes of Attachment Based Family Therapy (ABFT) as an aftercare model to further gains made in inpatient treatment and reduce risk factors for future suicide attempts.

DETAILED DESCRIPTION:
Annually, more adolescents and young adults in the United States die from suicide than from cancer, heart disease, AIDS, birth defects, stroke, pneumonia, influenza and chronic lung disease combined (U.S. Public Health Service, 1999). Each year approximately 1 in 5 teenagers seriously consider killing themselves, over one million teenagers attempt suicide, and between 1,600 and 2,000 die by suicide (U.S. Public Health Service, 1999). Clearly, the need for more empirically based treatment models is urgently needed.

Typically, after a suicide attempt or reporting of suicidal ideation with an intent or plan to kill themselves, adolescents are treated in a psychiatric hospital. In the past, an inpatient stay could provide intensive individual, group, family, and or medication therapy. However, managed care has shifted the goal of hospitalizations from treatment to stabilization. Adolescents are discharged when they are deemed to be no longer a threat to themselves, leaving the treatment of precipitating factors to outpatient aftercare. In a recent review of 21 studies on compliance with aftercare, Daniel and colleagues (2004) found that a majority of youth do received aftercare, but that noncompliance is very high. Very little evidence was found to support the effectiveness of aftercare. Surprisingly there are no studies on preventing adolescent reattempts of suicide after hospitalization. Important studies by Harrington et al. (1998) and King et al. (2007) have shown some promising results for aftercare reducing suicidal ideation, but no published studies have looked at preventing reattempts. Given the dearth of treatment studies for youth attempting suicide in general, it is not surprising that there are even fewer studies of aftercare for this population. Yet, given the high cost of even a short inpatient treatment, developing and testing effective aftercare programs that build on the gains made in inpatient treatment for youth who attempt suicide seems warranted.

One promising outpatient treatment approach for this population is Attachment-Based Family Therapy (ABFT; Diamond et al., 2002). ABFT is a manualized, brief (i.e., 12 to 16 week) family-based model designed specifically for treating depressed and suicidal adolescents. The model aims to reduce adolescent depression, suicidal ideation, family conflict, parental criticism, and adolescent isolation and hopelessness; all factors associated with adolescent suicide attempts (e.g., Brent et al., 1988). To accomplish these goals with the parent, ABFT aims to increase parental warmth, communication skills, and appropriate monitoring. For the adolescent, treatment aims to improve interpersonal problem solving, emotional regulation, and reengagement with positive prosocial activities (e.g., school, job, peers). As communication improves and trust is rebuilt, the parents reclaim their position as a secure base for adolescent development. The family becomes a context where adolescents learn to express their emotions and thoughts (including their suicidal ideation) in a differentiated and regulated manner, problem solve, and control their impulses. In many families, repairing the attachment rupture requires a "working through" of prior traumatic events (e.g., loss, divorce, abuse) often associated with the suicidal behavior. As adolescents become less preoccupied with suicide ideation and family conflict, treatment focuses on parents helping their adolescent navigate the challenges of school, peer relations and other life domains.

ABFT has recently proven effective in reducing suicidal ideation and depressive symptoms in a non-hospitalized population identified in primary care (Diamond et al., 2007). This grant will set the foundation for a programmatic look at treating adolescents who have been psychiatrically hospitalized for attempting suicide. This study will have two improvements over current aftercare services. First, it will improve the quality of aftercare by using an empirically based, family-based, manualized treatment. Second, it will rely on a continuity of care model where aftercare treatment begins while families are still in the hospital, potentially enhancing treatment compliance once the adolescent leaves the hospital.

* Objective 1: Develop a collaborative relationship with Belmont Psychiatric hospital and their Therapeutic Bridge Program to foster a research infrastructure that can support future adolescent suicide clinical trials research. This will include integrating standardized assessment tools into the inpatient procedures and establishing procedures for making referrals to the research program.
* Objective 2: Evaluate the feasibility and acceptability of ABFT outpatient aftercare for youth with a suicide attempt, after discharge from inpatient care. This will be evaluated by our ability to make contact with at least 80% of eligible patients, collect weekly follow up data, obtain at least 90% post treatment data, meet our recruitment goals, retain patients in treatment for at least 10 sessions, and be rated high on patient report of treatment acceptability and satisfaction.
* Objective 3: In an exploratory fashion, examine the differential effect sizes between Enhanced Usual Care (EUC) and ABFT at 14 weeks post hospital discharge for a) preventing future suicide attempts, b) reducing associated risk factors (suicide ideation, depression, and family conflict) and c) increasing treatment compliance (e.g., time to first session, number of sessions attended).

ELIGIBILITY:
Inclusion Criteria:

* in inpatient mental health treatment
* report a suicide attempt in the past month
* have a primary caretaker willing to participate in aftercare
* are able to travel to CHOP
* have no history of psychosis or low intellectual capacity
* speak adequate English.

Exclusion Criteria:

* being discharged to a residential placement

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ) | 14 weeks
  The CSQ is a 31 item questionnaire with responses on a 4-point scale. There are no subscales, and a total score is computed by summing scores across items. Higher scores indicate higher levels of satisfaction. In a variety of studies, the CSQ has demonstrated good internal consistency and predictive validity and has been reviewed favorably by several independent sources (Attkisson & Greenfield, 1994; Ogles et al., 2002). The CSQ has 8 items, and takes approximately 5 minutes to complete
Cornell Services Index (CSI) | baseline, 14 weeks
  The CSI is a self-report measure of medical and psychological services received (treatment utilization). We will complete information on type of provider, site of service, time to first session, and frequency of service, psychiatric assessments, pharmacotherapy, and individual and family therapy. The Cornell Services Index has been found to have good test-retest and interrater reliability. The Cornell has 32 items, and takes approximately 10 minutes to complete.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | baseline, weekly, 14 weeks
  The second edition of the BDI is a widely-used, 21-item self-report instrument designed to assess the severity of depressive symptoms in adults and adolescents. The BDI-II has high internal reliability (alpha = .91) and is highly and positively correlated with other measures of depression. The sensitivity and specificity for detecting depression in psychiatric patients has been established. With the original BDI, we found an alpha of .85 for 97 African American adolescents screened for a depression treatment pilot study. The BDI-II has 21 items, and takes approximately 5 minutes to complete.
Relatedness Scale (RS) | baseline, 14 weeks
  The relatedness scale is a 23-item measure assessing the relationships between children and their mother and father. There are two subscales: psychological proximity and emotional quality of the relationship. The psychological proximity seeking section of the measure has 12 statements each with a four point likert scale ranging from not at all true to very true. Similarly, the emotional quality section has 11 statements with a four-point response set ranging from almost never to almost always. The total score for the measure is the sum of the responses in each section.
Relationship Structures Questionnaire (RSQ) | Baseline, 14 weeks
  The RS is a self-report measure assessing attachment patterns in four domains: mother, father, romantic partner, and best friend. Each domain has ten items assessed on a 7-point likert scale ranging from strongly disagree to strongly agree. Each domain generates two scores: one for attachment related avoidance and the other for attachment related anxiety. The RS measures one component of attachment (i.e., avoidance and anxiety), which is a central change mechanism of ABFT.
Suicide Ideation Questionnaire (SIQ-JR) | baseline, weekly, 14 weeks
  The SIQ-JR is a 15-item version of the Suicidal Ideation Questionnaire. It is based on Reynolds' theoretical notion of suicidality forming a continuum ranging from thoughts of death, thoughts of wanting to be dead, general and specific suicidal plans, preparations for carrying out plans, and actual suicide attempts. It was originally designed for younger adolescents but has been frequently used in studies with older adolescents.
Columbia Suicide-Severity Scale (C-SSRS) | baseline, 14 weeks (if attempt made during treatment)
  The C-SSRS is an interview-based rating scale designed to create a topology of suicidal behavior and ideation. It assesses type of behavior, lethality of suicide attempts, and suicidal ideation, each scored as independent continuous measures. The C-SSRS is the prospective counterpart to the FDA suicide reclassification analysis and is currently being used in the National Institute of Mental Health (NIMH)funded multi-site trial, Treatment of Adolescent Suicide Attempters (TASA). The C-SSRS has 26 items
Suicide Intent Scale (SIS) | baseline, weekly and 14 week as needed
  The SIS is a 20-item, interviewer-administered assessment of the intensity of the attempter's wish to die at the time of the index attempt. Major constructs of the SIS have been found to be predictive both of future suicide attempts and suicide completions. The SIS has 20 items, and takes approximately 10 minutes to complete. The SIS is only given at the weekly and post treatment assessments if there has been a suicide attempt since the last assessment.
Lethality of Suicide Attempt Rating Scale | baseline, weekly and 14 weeks as needed
  Lethality of past suicide attempts will be assessed using this 11-item scale that assesses the medical lethality of attempts. The scale has high inter-rater reliability, excellent six-month test-retest reliability, and evidence of concurrent validity. The Lethality Scale has 7 items, and takes approximately 7 minutes to complete. The Lethality Scale is only given at the weekly and post treatment assessments if there has been a suicide attempt since the last assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Guy S. Diamond, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Diamond GS, Levy S. Bindungsorientierte Familientherapie als ambulante Nachsoge fur Jugendliche nach Suizidversuch. Psychotherapie im Dialog 13: 41-45, 2012.
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832